CLINICAL TRIAL: NCT06838754
Title: Effects of Whole Body Vibration on Gait Parameters and Postural Control in Children With Down Syndrome
Brief Title: Effect of Whole Body Vibration on Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/24/0716
Record Dates: First submitted 2024-11-03; First posted 2025-02-21 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Down Syndrome
Keywords: Down syndrome; Motor skills; Vibrations
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: It will be randomised control trial in which non probability snowball sampling will be used. Two groups of 5-12 age will be performed in which participants will be randomly divided. Group A will be receive Whole body Vibrations and routine physical therapy and Group B will be receive routine therapy.
Who Masked: Participant
Masking Description: Participants will receive separate treatment protocols and possible effects will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole body vibration therapy (Experimental): Experimental group will receive whole body vibrations while sitting. Walking in all directions,
  Interventions: Other: Whole body vibration therapy
- Routine physical therapy (Other): Group B will be the only one performing routine physical therapy (RPT). Stretching exercises will be part of these regular workouts. Walking in all directions,
  Interventions: Other: Routine physical therapy

INTERVENTIONS:
Other: Whole body vibration therapy — Experimental group will get whole body vibrations. WBV will be performed by the patient while seated on the vibrating plate's base. Five series with a 30-second wait will make up each session. Five minutes and thirty seconds will be spent on vibration, and twenty minutes and thirty seconds will be spent on exercise. 5 Hz will be the frequency utilized. Over the course of two months, 16 classes will be held twice a week.
  Arms: Whole body vibration therapy
Other: Routine physical therapy — Group B will only get routine physical therapy. Walking in all directions, advancing past the point of stability in a variety of positions, including half-kneeling, standing on both soft and hard surfaces, stepping up and down, walking and standing simultaneously, and standing on one leg with eyes open and closed were all part of the postural control exercise. There will be a 20-minute session.As each participant's functional improvement progresses, the intensity of the workout program will progressively rise. There will be 16 sessions in total (two days a week), with 8 sessions for each group.
  Arms: Routine physical therapy

SUMMARY:
A congenital condition known as Down syndrome is typified by an excess of genetic material from chromosome 21, making 47 chromosomes in total. Development of the body and brain may be impacted. About 1 in 700-1100 live births have the condition, and 1 in 700-1100 live births inherit it. Heart disease, hypotonia, ligament laxity, cerebral disabilities, thyroid abnormalities, and metabolic diseases are among the physical, cognitive, and metabolic changes that define it. Reduced performance, increased energy consumption, and altered gait patterns are frequently the results of motor disorders. This study intends to ascertain the effects of whole body vibrations (WBV), an activity that has been recommended for individuals with Down syndrome, on gait parameters and postural control in children with this condition.

DETAILED DESCRIPTION:
Whole Body Vibration (WBV) and routine physical therapy (RPT) are given to Group A, whereas routine physical therapy is given to Group B as a control. Two sessions of 20 minutes each are given to both groups twice a week. Postural control and gait metrics are the outcomes that will be examined. The present investigation will be conducted over a two-month period and will be a randomized control experiment. Alkhidmat Hospital in Sargodha and Al-Ghafoor Hospital in Bhera will provide the data. 16 participants will participate in the trial; they will be randomly assigned to two equal groups. Children with DS, ages 5 to 12, of both sexes, will be eligible to participate in the study. The condition of improved comprehension of children older than five years was taken into consideration when determining the inclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Ages 5-12
* Both sexes are chosen
* Children with Down syndrome older than 5 who are more knowledgeable about the exercise to be done are given preference.

Exclusion Criteria:

* Children with cardiac conditions and other conditions
* Atlantoaxial instability and prosthesis implantation are excluded.
* DS kids who don't have their parents or legal guardians sign the consent form.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-02-23 (Actual); Study Completion 2025-03-07 (Actual)

PRIMARY OUTCOMES:
Step length | 2 months.
  Step length will be measured from consecutive heel contacts in cm.
Posture and postural ability test (PPAS) | 2 months.
  The PPAS assesses 4 positions. Standing, sitting, supine and prone Each position is assessed according to the postural ability, quality of posture and within postural ability seven levels are designated, ranging from Level 1 = 'Unplaceable in an aligned posture' to 7 = Able to move into and out of position.
Stride length | 2 months.
  Stride length is the distance between the previous heel strike of the right foot and the new heel strike of the right foot and measured in cm.
Step width | 2 months.
  Step width will be measured from the mediolateral space between the two feet in cm.
Foot angle | 2 months.
  Foot angle will be measured by the angle between the line of progression and the foot axis in degree.

CONTACTS AND LOCATIONS:
Overall Officials: Tuba Sameen, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yaqoob M, Manzoor J, Hyder SN, Sadiq M. Congenital heart disease and thyroid dysfunction in Down syndrome reported at Children;s Hospital, Lahore, Pakistan. Turk J Pediatr. 2019;61(6):915-924. doi: 10.24953/turkjped.2019.06.013. PMID 32134586